CLINICAL TRIAL: NCT05859633
Title: Neutrophil/Lymphocyte Ratio in Predicting the Severity of Acute Pancreatitis
Brief Title: Neutrophil/Lymphocyte Ratio in Acute Pancreatitis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Romany Waheed Morkis Beshay, Internal Medicine, Assiut University
Other Study IDs: Romay
Record Dates: First submitted 2023-05-04; First posted 2023-05-16 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2023-05

CONDITIONS: Acute Pancreatitis
MeSH Terms: conditions — Pancreatitis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients with acute pancreatitis: any patient suffers from acute pancreatitis
  Interventions: Diagnostic Test: Neutrophil/Lymphocyte Ratio in acute pancreatitis

INTERVENTIONS:
Diagnostic Test: Neutrophil/Lymphocyte Ratio in acute pancreatitis — role of Neutrophil/Lymphocyte Ratio in acute pancreatitis

SUMMARY:
Acute pancreatitis (AP) is a disease characterized by dysfunction of pancreatic acinar cells, improper activation of trypsin, and subsequent destruction of pancreatic self-defense mechanisms, further exacerbating injury and damage of pancreatic cells. It is a rapidly developing inflammatory process of the pancreas, and the most common reasons are alcohol and gallstones.

DETAILED DESCRIPTION:
As one of the most common gastrointestinal diseases in hospitalized patients, the incidence of AP has gradually increased and is 4.9 to 73.4 cases per 100,000 people worldwide in the past few decades, imposing a heavy burden on the health system and leading to long-term hospitalization, most medical costs, and significant mortality.

Up to 10% to 20% of AP patients will develop SAP, and the leading cause of poor prognosis in patients with AP is a vital organ (cardiovascular organs, lung, and kidney) failure and pancreatic necrosis . In clinical practice, varieties of scoring systems are available and have been gradually confirmed, such as the Ranson score, Glasgow score, Acute Physiology and Chronic Health Evaluation (APACHE II), BISAP, and computed tomography severity index (CTSI) . These systems are cumbersome and take a long time to operate, requiring a lot of parameters that are not routinely collected in the early stages of the disease. For example, the BISAP score is characterized by high specificity, but its sensitivity to SAP is not satisfied. Therefore, their early prediction power is not good.

In AP, inflammation first activates a series of inflammatory cytokines, proteolytic enzymes, and anaerobic radioactive nucleic acids to destroy the tissue. The degree of neutrophils decrease is related to the improvement of prognosis of AP, while the degree of lymphocyte increase is related to the severity of the disease. The neutrophil-lymphocyte ratio (NLR) is a more comprehensive biomarker that used neutrophil and lymphocyte counts to respond rapidly to the extent of inflammatory progression and serves as a useful predictive marker to identify the severity of AP. It is well known that AP is a fast-onset inflammation of the pancreas, and an effective prediction of the severity of AP can guide AP patients to receive adequate treatment earlier, contributing to a better prognosis.

ELIGIBILITY:
Inclusion Criteria:

* patients with acute pancreatitis

Exclusion Criteria:

* Patients with acute abdomen with diagnosis other than AP
* Patients with AP who are under age of 18 years old
* Patient's refusal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any patient who is above age of 18 years old and diagnosed to have AP. Patients were diagnosed with acute pancreatitis if more than 2 of the following conditions were satisfied: 1) abdominal pain consistent with acute pancreatitis (acute onset of a persistent, severe, epigastric pain often radiating to the back); 2) serum amylase and/or lipase level at least 3 times greater than the upper limit of the normal value; and 3) characteristic manifestation of acute pancreatitis on contrast-enhanced computed tomography, magnetic resonance imaging, or transabdominal ultrasonography
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-05-30 (Estimated); Primary Completion 2023-12-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
severe acute pancreatitis | one year
  frequency of severe acute pancreatitis

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed M Abu-Elfatth, Principal Investigator — Assiut University
Locations (1):
- Ahmed Mohammed Abu-Elfatth, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
undecided

REFERENCES:
- [Background] Mederos MA, Reber HA, Girgis MD. Acute Pancreatitis: A Review. JAMA. 2021 Jan 26;325(4):382-390. doi: 10.1001/jama.2020.20317. PMID 33496779